CLINICAL TRIAL: NCT06890338
Title: A Single-Arm, Phase 2 Study of Neoadjuvant Carboplatin and Mirvetuximab Soravtansine in Subjects With FRα-Expressing Advanced-Stage Serous Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: A Study to Assess Anti-Tumor Activity of Intravenously (IV) Infused Carboplatin With Mirvetuximab Soravtansine in Participants With Newly Diagnosed Folate Receptor Alpha (FRα)Expressing Advanced-Stage Serous Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M25-231; GOG-3115 (Other: GOG)
Record Dates: First submitted 2025-03-20; First posted 2025-03-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer; Neoadjuvant
Keywords: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer; Neoadjuvant; Interval Debulking Surgery; Mirvetuximab Soravtansine; MIRV; IMGN853; ELAHERE(R); Carboplatin; Bevacizumab
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — Carboplatin; mirvetuximab soravtansine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Carboplatin + Mirvetuximab Soravtansine (Experimental): Participants will receive carboplatin in combination with mirvetuximab soravtansine on Day 1 of a 21-day cycle per dose +/- Bevacizumab per investigator's discretion.
  Interventions: Drug: Carboplatin; Drug: Mirvetuximab Soravtansine; Drug: Bevacizumab

INTERVENTIONS:
Drug: Carboplatin — Intravenous (IV) infusion
Drug: Mirvetuximab Soravtansine — Intravenous (IV) infusion
  Other Names: MIRV; IMGN853; ELAHERE™
Drug: Bevacizumab — Intravenous (IV) infusion (per investigator's discretion)

SUMMARY:
Cancer is a condition where cells in a specific part of body grow and reproduce uncontrollably. The purpose of this study is to assess the safety and efficacy of neoadjuvant carboplatin and mirvetuximab soravtansine in participants with folate receptor alpha (FRα) -expressing advanced-stage serous epithelial ovarian, fallopian tube or primary peritoneal cancer (EOC).

Mirvetuximab Soravtansine (MIRV) is an investigational antibody drug conjugate designed to selectively kill cancer cells. The antibody (protein) part of MIRV targets tumors by delivering a cell-killing drug to cancer cells carrying a protein called folate receptor alpha (FRα). This is a single arm study in adult participants with advanced-stage Fédération Internationale de Gynécologie et d'Obstétrique (FIGO) III-IV FRα-expressing serous EOC. Around 140 participants will be enrolled in the study at approximately 80 sites in the United States.

Participants will receive intravenous infusion of MIRV in combination with carboplatin on day 1 of each cycle, every 21 days for up to 6 - 9 Cycles. The total study duration will be approximately 3 years .

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic and may require frequent medical assessments, blood tests, and scans.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Be judged by the investigator and/or treating physician to be an appropriate candidate to receive neoadjuvant chemotherapy.
* Diagnosis of biopsy-confirmed high-grade, serous epithelial ovarian, fallopian tube or primary peritoneal cancer.
* Participant meets the following disease criteria:

  * Stage III or IV disease by the Fédération Internationale de Gynécologie et d'Obstétrique (FIGO) staging system, 27 and
  * Folate Receptor Alpha (FRα) expression positivity as defined by immunohistochemical staining of >= 75% of viable tumor cells with moderate (2+) and/or strong (3+) membrane staining by the AbbVie specified vendor with the Ventana Folate Receptor Alpha (FOLR1) assay, and
  * Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 criteria.

Exclusion Criteria:

* Endometrioid, clear cell, mucinous, or sarcomatous tumor histology; mixed tumors containing any of the above histologies; or low-grade/borderline ovarian tumor.
* Previous clinical diagnosis of noninfectious interstitial lung disease, including noninfectious pneumonitis.
* Previously treated with anticancer therapy including chemotherapy, radiation therapy, immunotherapy, or biologic agent for current cancer, with the exception of one cycle of single agent carboplatin
* Participants with the following ocular history and/or concurrent disorders:

  * History of corneal transplantation;
  * Undergoing active postoperative management for refractive surgery, cataract surgery, corneal cross-linking, or corneal complications of surgery;
  * Confluent superficial punctate keratopathy (SPK) not expected to resolve to non-confluence or better within the screening window with standard of care (SOC) intervention;
  * Active or chronic clinically significant (>= Grade 3) corneal dystrophy (e.g., Fuchs dystrophy);
  * Active ocular conditions requiring ongoing treatment/monitoring, such as glaucoma, which is not adequately controlled with medication or surgery, wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, macular degeneration, presence of papilledema or an ocular condition with high risk of retinal detachment;
  * Monocular vision with visual acuity in the worse eye, worse than 20/200 or visual fields less than 20 degrees (i.e., functional blindness in at least one eye).
* History of other malignancy within 3 years prior to signing study consent. -- Note: Participants with tumors with a negligible risk for metastasis or death (e.g., adequately controlled basal-cell carcinoma or squamous-cell carcinoma of the skin, or carcinoma in situ of the cervix or breast) are eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Objective Response (OR) by Independent Central Review (ICR) | Up to Approximately 3 years
  OR is defined as the best overall response of radiographic complete response (CR) or partial response (PR) as assessed by ICR using RECIST Version 1.1 criteria, prior to any subsequent anticancer therapy, including interval debulking surgery (IDS).

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events (AE) | Up to Approximately 3 years
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with the treatment. The investigator assesses the relationship of each event to the use of study drug.
Percentage of Participants with AEs leading to study drug discontinuation or dose modification | Up to Approximately 3 years
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with the treatment. The investigator assesses the relationship of each event to the use of study drug.
Objective Response (OR) by Investigator | Up to Approximately 3 years
  Or is defined as the best overall response of radiographic CR or PR as assessed by investigator using RECIST Version 1.1 criteria, prior to any subsequent anticancer therapy, including IDS.
Disease Control by ICR | Up to Approximately 3 years
  Disease control defined as CR, PR, or stable disease (SD) as assessed by ICR per RECIST Version 1.1 prior to subsequent anticancer therapy including IDS.
Disease control by Investigator | Up to Approximately 3 years
  Disease control defined as CR, PR, or stable disease (SD) as assessed by investigator per RECIST Version 1.1 prior to subsequent anticancer therapy including IDS.
Percentage of Participants With CA-125 Confirmed Response Per Gynecologic Cancer Intergroup (GCIG) Criteria | Up to Approximately 3 years
  The GCIG CA-125 response was defined as at least 50% reduction in CA-125.
Progression-Free Survival (PFS) as assessed by investigator | Up to Approximately 3 years
  PFS as assessed by investigator per RECIST v1.1 is defined as the time from the date of C1D1 until investigator-assessed PD or death (whichever occurs first).
Percentage of Participants that Underwent Interval debulking surgery (IDS) | Up to Approximately 3 years
  Percentage of participants that underwent IDS during the course of the study treatment
Percentage of participants with Grossly complete tumor cytoreduction at IDS | Up to Approximately 3 years
  Grossly complete tumor cytoreduction is defined as the absence of macroscopically visible residual disease at the end of the surgery
Percentage of participants with Near-Complete Tumor Cytoreduction at IDS | Up to Approximately 3 years
  Defined as macroscopically visible residual tumor ≤ 1 cm at the end of surgery.
Time to deterioration in disease-related symptoms as measured by the NCCN-FACT Ovarian Symptom Index (NFOSI-18) disease symptom subscale - physical (DRS-P) | Up to Approximately 3 years
  The NFOSI-18 provides a total score that sums all 18 items, plus 2 multi-item scales that assess physical disease-related symptoms (DRS-P; 9 items) and general function/well-being (F/WB; 3 items).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (46):
- United States (46):
  - University of Alabama at Birmingham (UAB) Hospital /ID# 274793, Birmingham, Alabama
  - Usa Mitchell Cancer Institute /ID# 276022, Mobile, Alabama
  - California Pacific Medical Center /ID# 275329, San Francisco, California
  - Ridley Tree Cancer Center /ID# 275219, Santa Barbara, California
  - Danbury Hospital, Western Connecticut Health Network /ID# 274783, Danbury, Connecticut
  - Norwalk Hospital /ID# 274561, Norwalk, Connecticut
  - Jupiter Medical Center /ID# 276616, Jupiter, Florida
  - Mount Sinai Medical Center /ID# 274868, Miami, Florida
  - OSF St. Francis Medical Center /ID# 274752, Peoria, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center /ID# 275492, Indianapolis, Indiana
  - Baptist Health Lexington /ID# 275218, Lexington, Kentucky
  - Women'S Cancer Care /ID# 276469, Covington, Louisiana
  - University Medical Center New Orleans /ID# 274755, New Orleans, Louisiana
  - Trials 365 /ID# 274310, Shreveport, Louisiana
  - Holy Cross Hospital /ID# 275872, Silver Spring, Maryland
  - Metro Minnesota Community Oncology Research Consortium (MMCORC) /ID# 274780, Saint Louis Park, Minnesota
  - Cox Medical Center South /ID# 274826, Springfield, Missouri
  - The Center Of Hope /ID# 274313, Reno, Nevada
  - Rutgers Cancer Institute of New Jersey /ID# 274358, New Brunswick, New Jersey
  - Holy Name Medical Center /ID# 276240, Teaneck, New Jersey
  - Optimum Clinical Research Group /ID# 274583, Albuquerque, New Mexico
  - Imbert Cancer Center /ID# 275634, Bay Shore, New York
  - Northwell Health Cancer Institute At Huntington /ID# 276814, Greenlawn, New York
  - Northwell Health Center for Advanced Medicine. /ID# 275641, Lake Success, New York
  - Northwell Health Queens Cancer Center /ID# 274850, Rego Park, New York
  - University of North Carolina Medical Center /ID# 275307, Chapel Hill, North Carolina
  - Sanford Fargo Medical Center - Fargo /ID# 275489, Fargo, North Dakota
  - The Mark H Zangmeister Center /ID# 275106, Columbus, Ohio
  - Oncology Associates of Oregon, P.C. /ID# 275006, Eugene, Oregon
  - Northwest Cancer Specialists /ID# 275101, Portland, Oregon
  - St. Lukes University Hospital /ID# 274362, Bethlehem, Pennsylvania
  - University of Pennsylvania /ID# 275612, Philadelphia, Pennsylvania
  - Women & Infants Hospital /ID# 274716, Providence, Rhode Island
  - Sanford Cancer Center /ID# 274901, Sioux Falls, South Dakota
  - Avera Cancer Institute - Sioux Falls /ID# 276226, Sioux Falls, South Dakota
  - Texas Oncology - Austin Central /ID# 275046, Austin, Texas
  - Texas Oncology - Fort Worth Cancer Center /ID# 275043, Fort Worth, Texas
  - Houston Methodist Hospital /ID# 274568, Houston, Texas
  - Texas Oncology - San Antonio Medical Center - Research Drive /ID# 275090, San Antonio, Texas
  - Texas Oncology - The Woodlands /ID# 275015, The Woodlands, Texas
  - Texas Oncology - Northeast Texas /ID# 275057, Tyler, Texas
  - UVA Health University Hospital /ID# 275309, Charlottesville, Virginia
  - Inova Schar Cancer Institute - Fairfax - Innovation Park Drive /ID# 276456, Fairfax, Virginia
  - Carilion Clinic /ID# 274684, Roanoke, Virginia
  - Providence Sacred Heart Medical Center & Children'S Hospital /ID# 274585, Spokane, Washington
  - West Virginia University School of Medicine /ID# 274556, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-231